CLINICAL TRIAL: NCT06643364
Title: The Effects of Vision Training Applied to Kumite Karate National Team Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Tuğba Kuru Çolak, Principal İnvestigator (Professor Doctor), Marmara University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MU-SBE-FTR-MŞE-02
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Health Individuals; Atlhetes
Keywords: vision training; vision acuity; reaction time

STUDY DESIGN:
Intervention Model Description: There are two groups: one group is the control group and the other is the vision training group, in which vision training is applied
Who Masked: Investigator, Outcomes Assessor
Masking Description: All athletes who participated in the study, the researcher who performed the measurements and the people who performed the statistical evaluation did not know which athlete was in which group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): The karate athletes in the control group continued their routine training planned by the national team during the study.
  Interventions: Other: Routine Training Program
- Vision Training Group (Experimental): The karate athletes in the vision training group participated in a vision training programme that included eye movements and was applied by one of the researcher physiotherapists in addition to their routine training planned by the national team. The application was applied for 10 minutes in 3 sessions per week for 4 weeks.
  Interventions: Other: Vision Training Program; Other: Routine Training Program

INTERVENTIONS:
Other: Vision Training Program — Vision Training Programme: A training programme including exercises such as saccadic movements of the eye, spiral movements, converging-diverging exercises, peripheral walking was applied.
  Arms: Vision Training Group
Other: Routine Training Program — All athletes continued their routine training programmes planned by the national team coaches for karate sport during the training period.

SUMMARY:
This study examines the effects of visual training applied to professional kumite karate athletes. In karate, rapid decision-making, opponent perception at the right time, effective implementation of strategic moves and reaction time are largely dependent on visual perception skills. In this context, our study investigated how vision training improves visual acuity and sportive performance of kumite karate athletes.

DETAILED DESCRIPTION:
Before the study, ethical approval was obtained from Marmara University Faculty of Medicine Ethics Committee with the number 09.2024.611. The study was started with 24 national athletes from Kocaeli Metropolitan Municipality Kağıtspor Team and was carried out on 23 athletes after one athlete in the control group was injured. The athletes who were examined by an ophthalmologist before the study, who did not have any visual problems and who did not have any surgical operation and/or injury history that would adversely affect the balance in the last 6 months were randomly divided into 2 groups. The 12-member vision training group was subjected to a vision training programme that included eye exercises accompanied by a physiotherapist for 3 sessions per week in addition to their routine training for 4 weeks, while the control group continued their routine training. At the beginning of the study (week 0) and at the end of the training (week 4), 't ruler-nelson hand reaction test', 'sit & lie flexibility test' were performed by another physiotherapist, and 'snellen test' measurements were performed by an ophthalmologist for 'visual acuity' evaluation of the athletes. The researcher who performed the reaction time and flexibility measurements and the physician who assessed visual acuity performed the measurements without knowing which group the athletes were in. After statistically homogeneous-normality evaluation of the groups, Independent Sample t Test was used for comparison of descriptive characteristics between the groups. Mixed-order analysis of variance (ANOVA) was used to compare the variables in the groups according to the follow-up times. Bonferroni correction was applied for the comparison of main effects in the analyses. p<0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Being a 'Karate-Do' style athlete in Kocaeli Metropolitan Municipality Kağıtspor
* To be at A national team level
* To continue active sports life
* To be between the ages of 15-35

Exclusion Criteria:

* Having any eye disease
* Any surgery or serious pathology in the last 6 months
* Any history of traumatic brain injury in the last 6 months
* Upper/lower extremity injury in the last 3 months
* Having one of the systemic disorders (such as musculoskeletal system, respiratory system) Being younger than fifteen years old and older than thirty-five years old History of a disease related to balance, vestibular system Regular use of medication related to the vestibular system, vision and balance Presence of congenital anomalies

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2024-07-16 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2024-10-08 (Actual)

PRIMARY OUTCOMES:
Visual Acuity Assessment | Pre-study (week 0) and post-study (week 4)
  Visual acuity was assessed by an ophthalmologist using a Snellen chart.

SECONDARY OUTCOMES:
Reaction Time Assessment (cm) | Pre-study (week 0) and post-study (week 4)
  It is a test that measures reaction time to visual stimuli. In the hand reaction test, the ruler is placed between the fingers of the hand. The practitioner holds the ruler by the tip and above. He/she releases the ruler a while after giving the ready signal. The subject tries to catch the ruler as soon as possible. The reaction time is calculated and recorded according to the distance at the point of catching. 3 repetitions are done and the average value is recorded.
Sit & Reach Test (cm) | Pre-study (week 0) and post-study (week 4)
  Sit on the floor and rest bare feet flat on the test bench. The torso (waist and hips) is tilted forward and the knees are asked to reach as far as possible forward without bending the knees, with the hands in front of the body. The subject tries to reach the farthest point in this way and waits 2 seconds at the last point and the value is recorded. The tester stands next to the subject and prevents the subject's knees from bending. The test is repeated three times and the average value is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Tugba KURU COLAK, Prof.Dr., Study Director — Marmara University
Locations (1):
- Kocaeli Metropolitan Municipality Kağıtspor, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No